CLINICAL TRIAL: NCT06520475
Title: Efficacy of Bupivacaine-magnesium Combination Versus Bupivacaine Alone in Genicular Nerve Block in Total Knee Replacement Surgeries: a Randomized Controlled Study
Brief Title: Efficacy of Bupivacaine-magnesium Combination Versus Bupivacaine Alone in Genicular Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-157-2024
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine + Magnesium (Active Comparator)
  Interventions: Procedure: genicular nerve block using bupivacaine and magnesium
- Bupivacaine + Normal saline (Placebo Comparator)
  Interventions: Procedure: genicular nerve block using bupivacaine and normal saline

INTERVENTIONS:
Procedure: genicular nerve block using bupivacaine and magnesium — The patients will receive 13 ml of 0.5% bupivacaine and 2 ml of 10% magnesium sulfate
  Arms: Bupivacaine + Magnesium
Procedure: genicular nerve block using bupivacaine and normal saline — The patients will receive 13 ml of 0.5% bupivacaine and 2 ml of normal saline
  Arms: Bupivacaine + Normal saline

SUMMARY:
It is proved that the addition of magnesium sulfate to local anesthetics for neuraxial anesthesia improves the quality of analgesia and prolongs the duration of anesthesia . In-vitro and in-vivo studies have demonstrated that magnesium enhances the local anesthetics effect on peripheral nerves .

No previous studies were conducted on magnesium sulfate as an adjuvant to the local anesthetic in genicular nerve block. Hence, this study will be conducted to assess analgesic efficacy of magnesium sulfate when added to bupivacaine in ultrasound guided genicular nerve block

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) I or II physical status.
* Between 18 and 70 years of age.
* Both genders.
* Patients undergoing total knee replacement surgery.

Exclusion Criteria:

* Patient refusal.
* ASA Ⅲ and Ⅳ patients.
* Known allergy to the study drugs.
* Hypermagnesemia.
* Central or peripheral neurological disease.
* Pregnancy.
* Drug or alcohol abuse.
* Localized infection at the site of the block.
* Bleeding disorder (platelets count less than 100,000 or international normalized ratio more than 1.4)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 24 hours post-operatively
  Pain will be assessed with Numerical Rating Scale. Patients will be asked to circle the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible.

SECONDARY OUTCOMES:
First request for analgesia | 24 hours post-operatively
Total opioid consumption | 24 hours post-operatively
Patient satisfaction | 24 hours post-operatively
  Patient satisfaction will be assessed at 48 h postoperatively (0 = very dissatisfied, 2 = somewhat dissatisfied, 3 = somewhat satisfied, 4 = very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini hospital, Cairo, Egypt